CLINICAL TRIAL: NCT06400238
Title: MATCH Treatment Subprotocol Z1H: Phase II Study of Copanlisib in Patients With Tumors With Deleterious PTEN Sequencing Result and PTEN Expression by IHC
Brief Title: Testing Copanlisib as Potentially Targeting Treatment in Cancers With PTEN Expression (MATCH - Subprotocol Z1H)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-01162; NCI-2024-01162 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-Z1H (Other: ECOG-ACRIN Cancer Research Group); EAY131-Z1H (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-05-03; First posted 2024-05-06 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — Biopsy; Specimen Handling; copanlisib; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (copanlisib) (Experimental): Patients receive copanlisib IV over 60 minutes on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT or MRI during screening and on study, as well as during follow-up as clinically necessary. Patients undergo biopsies and blood sample collection on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Copanlisib; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Copanlisib — Given IV
  Other Names: BAY 80 6946; BAY 80-6946; BAY 806946; BAY-80-6946; BAY806946; PI3K Inhibitor BAY 80-6946
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This phase II MATCH treatment trial tests how well copanlisib works in treating patients with cancer that has certain genetic changes. Copanlisib is used in patients whose cancer has a mutated (changed) form of a gene called PTEN. It is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal protein that signals cancer cells to multiply. This helps slow or stop the spread of cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive copanlisib intravenously (IV) over 60 minutes on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) during screening and on study, as well as during follow-up as clinically necessary. Patients undergo biopsies and blood sample collection on study.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 1 year.

THE MATCH SCREENING TRIAL:

Please see NCT02465060 for information on the MATCH Screening Protocol and applicable documents.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol EAY131/ NCI-2015-00054 prior to registration to treatment subprotocol
* Patients must fulfill all eligibility criteria of MATCH Master Protocol at the time of registration to treatment step (Step 1, 3, 5, 7)
* Patients must have mutations in the PTEN gene with 1% or more expression of PTEN by immunohistochemistry (IHC) as determined via the MATCH Master Protocol

  * NOTE: For patients entering the study, all patients must have PTEN IHC performed as described in the MATCH Master Protocol. This includes patients entering the study via the outside assay process
* Patients must not have co-existing aberrations in the MAPK or PI3K/MTOR pathways as determined by the MATCH screening assessment in NRAS, HRAS, KRAS, BRAF, PIK3CA, AKT or mTOR
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients must not have known hypersensitivity to copanlisib or compounds of similar chemical or biologic composition
* Patients must not have had prior treatment with copanlisib or other PI3K inhibitors, AKT inhibitors or mTOR inhibitors
* Patients must not be on strong inhibitors or inducers of CYP3A4 within two weeks prior to start of study treatment and for the duration of study treatment
* Patients should stop using herbal medications at least 7 days prior to the first dose of copanlisib. Herbal medications include, but are not limited to: St. John's wort, kava, ephedra, gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, black cohosh and ginseng
* Patients with type I or II diabetes mellitus must have a glycosylated hemoglobin (HbA1c) ≤ 8.5% within 28 days from registration
* Patients must not have uncontrolled hypertension defined as systolic blood pressure (SBP) greater than 160 mmHg or diastolic blood pressure (BP) greater than 100 mmHg or use of more than 2 anti-hypertensive medications
* Patients must not have HER2 positive (3+ by IHC or fluorescence in situ hybridization [FISH] ratio ≥ 2) breast cancer
* Patients must not have indolent NHL (non-Hodgkin's lymphoma) or DLBCL (diffuse large B cell lymphoma) because other studies are ongoing with this agent in this group of patients
* Patients must not be on anti-arrhythmic therapy other than digoxin or beta-blockers
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9 /L
* Platelets ≥ 100 x10^9 /L
* Hemoglobin (Hb) > 9 g/dl
* Total serum bilirubin < 2.0 mg/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5x upper limit of normal (ULN) (< 5 x ULN in patients with liver metastases)
* Serum creatinine < 1.5 x ULN
* Patients with non-healing wound, ulcer, or bone fracture are not eligible
* Patients with history of or current interstitial pneumonitis are not eligible

  * NOTE: For solid tumors, cytomegalovirus (CMV) polymerase chain reaction (PCR) can be obtained at the discretion of treating physician or local institutional guidelines
* Men and women of child-bearing potential must agree to use contraception while receiving study treatment and for 1 month after the last dose of copanlisib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Filip Janku, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol Z1H was activated on June 20, 2018. Thirty-five patients were enrolled between October 2018 and January 2020. All patients were enrolled through the outside laboratory.
Pre-assignment Details: The PTEN mutation status was determined by a CLIA-approved assay performed in NCI-MATCH approved laboratory for all patients in this arm. Thirty-one out of the 35 outside lab patients had their samples centrally confirmed.
Groups:
- Treatment (Copanlisib): Patients receive copanlisib 60 mg IV over 60 minutes on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT or MRI during screening and on study, as well as during follow-up as clinically necessary. Patients undergo biopsies and blood sample collection on study.
Period: Overall Study
Arm/Group | Treatment (Copanlisib)
Started | 35
Started Protocol Therapy | 33
Eligible, Treated and Mutation Status Confirmed (Primary efficacy analysis set) | 29
Completed | 0
Not Completed | 35
Not completed — Started Protocol Therapy | 2
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Disease Progression | 27
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: Patients who were eligible, started protocol therapy, and had mutation status confirmed at the analysis time were the analyzable patients
Arm/Group | Treatment (Copanlisib)
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 59 [22 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Details about how to define complete response and partial response can be found in the master protocol. 90% two-sided binomial exact confidence interval is calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Copanlisib)
Number analyzed (Participants) | 29
percentage of participants | 3.4 [0.2 to 15.3]

2. Secondary Outcome: 6-month Progression Free Survival (PFS)
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS rate is determined
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Copanlisib)
Number analyzed (Participants) | 29
percentage of participants | 15.4 [6.1 to 28.7]

3. Secondary Outcome: Progression Free Survival
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Copanlisib)
Number analyzed (Participants) | 29
months | 1.84 [1.77 to 2.07]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All patients enrolled were included in the all-cause mortality analysis. Thirty-three patients were included in the toxicity analysis (excluding 2 who did not receive treatment).
Arm/Group | Treatment (Copanlisib)
All-Cause Mortality (participants affected / at risk) | 31/35
Serious Adverse Events (participants affected / at risk) | 16/33
Other Adverse Events (participants affected / at risk) | 27/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Copanlisib) (N=33)
Fatigue (General disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Soft tissue necrosis upper limb (Musculoskeletal and connective tissue disorders) | 1
Hypertension (Vascular disorders) | 6
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Copanlisib) (N=33)
Anemia (Blood and lymphatic system disorders) | 8
Chills (General disorders) | 3
Fatigue (General disorders) | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 16
Oral dysesthesia (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
Skin infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 5
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 13
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 4
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 5
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT06400238/Prot_000.pdf
  • Informed Consent Form (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT06400238/ICF_001.pdf